CLINICAL TRIAL: NCT06648187
Title: The Efficacy of Early Motor-Cognitive Integrative Training on Cognitive and Motor Performance in Patients With Aneurysmal Subarachnoid Hemorrhage: A Pilot Study
Brief Title: Early Motor-Cognitive Integrative Training on Cognitive and Motor Performance in Aneurysmal Subarachnoid Hemorrhage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202405012RINB
Record Dates: First submitted 2024-10-13; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Subarachnoid Aneurysm Hemorrhage
Keywords: Aneurysmal Subarachnoid Hemorrhage; Motor-Cognitive Integrative Training; Cognition; Early mobilization
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early motor-cognitive integrative training (e-MCIT) (Experimental): Evaluation will be conducted at three assessment time points including baseline assessment (following initial medical intervention), assessment at the time of discharge from the intensive care center (an average of 2 weeks), and discharge from the hospital (an average of 4 weeks). After recruiting in this study, participants all receive the intervention of e-MCIT.
  Interventions: Other: Early motor-cognitive integrative training (e-MCIT)

INTERVENTIONS:
Other: Early motor-cognitive integrative training (e-MCIT) — Early motor-cognitive integrative training (e-MCIT) is an approach where motor and cognitive training are conducted simultaneously. The intervention consists of 30-minute sessions, conducted 4-5 times per week, until discharging from the hospital. Both motor and cognitive training have five stages each, and their progression is independent, meaning that during training, a participant might be in the fourth stage of motor training and the second stage of cognitive training. According to hospital's policy, occupational therapy and speech therapy will be provided in schedule if needed. Motor training is derived from a previous protocol of early mobilization intervention applied to a population with SAH, which based on the ICU Mobility Scale. The activities of cognitive training target areas such as attention, orientation, language ability, memory, calculation, judgment, working memory, executive function, and daily living functions.

SUMMARY:
Despite its lower incidence rate within the stroke population and tendency to affect younger individuals, SAH carries the highest risk of PSCI. The neural mechanisms underlying these cognitive deficits remain poorly understood, but potential factors include treatment approaches, underlying disease pathophysiology, post-disease complications, or alterations in neural connectivity. Previous literature indicates that cognitive deficits in SAH primarily manifest in areas such as visuospatial skill, verbal memory language abilities (including verbal comprehension, verbal fluency, abstract language), executive function (working memory) and attention. These impairments significantly impact patients' ability to perform ADL independently and return to work, despite motor function recovery. This pilot study tests the feasibility, logistics, and methodology of the research project, as well as to identify any potential problems or challenges that may arise. In the future, the investigators plan to examine the impact of early intervention with MCIT (e-MCIT) on cognitive function, motor recovery, functional abilities, and ADL in acute SAH patients upon discharge from the ICU and during the post-intervention assessment. The hypothesis of this study is that there is feasibility and safety in early intervention with MCIT (e-MCIT) in aSAH patients. Otherwise, e-MCIT will result in significant improvements in cognitive function, motor recovery, functional abilities, and ADL among SAH patients upon discharge from the ICU and the post-intervention assessment (in future work will identify by comparing with early mobilization group only).

DETAILED DESCRIPTION:
Background and literature review: Spontaneous subarachnoid hemorrhage (SAH), often resulting from intracerebral aneurysm rupture is a relatively uncommon but impactful form of stroke predominantly affecting middle-aged individuals. Aneurysmal SAH (aSAH) presents a high risk of post-stroke cognitive impairment (PSCI) compared to other stroke types, with an occurrence rate ranging from 26% to 43%. Cognitive impairments, particularly in executive function, attention, memory, and language abilities, are prevalent among aSAH survivors, with notable differences observed in cognitive outcomes based on medical interventions such as clipping or coiling. Additionally, cerebral changes following aSAH, including delayed onset cerebral infraction, white matter hyperintensities and focal encephalomalacia, contribute to cognitive deficits. In clinical settings, patients with aSAH often demonstrate notable improvements in motor function recovery, however, cognitive issues, such as executive function and complex attention, are closely linked to patients' inability to perform the activities of daily living (ADL) independently and return to work, even after disease recovery. While physical therapy interventions, including early mobilization, show promise in enhancing functional outcomes, there is a dearth of research specifically addressing cognitive rehabilitation in aSAH patients.

Integration of motor-cognitive training approaches, such as motor-cognitive integrative training (MCIT), may hold potential for improving cognitive and motor recovery in SAH patients, akin to their application in other neurological disorders like Parkinson's disease and stroke. Understanding the intricate relationship between cognitive deficits and functional outcomes is crucial for developing targeted rehabilitation strategies to improve the quality of life for aSAH survivors.

Purpose: This pilot study tests the feasibility, logistics, and methodology of the research project, as well as to identify any potential problems or challenges that may arise. In the future, the investigators plan to examine the impact of early intervention with MCIT (e-MCIT) on cognitive function, motor recovery, functional abilities, and ADL in acute SAH patients upon discharge from the ICU and during the post-intervention assessment.

Study design: This is a pilot study to testify the feasibility, logistics, and methodology of evaluation and early motor-cognitive integrative training (e- MCIT) on cognitive function, motor recovery, functional ability and abilities in ADL in patients with aSAH in acute phase. The intervention commences during the acute setting in the ICU period and extends through the subacute phase in the hospital's general ward. Evaluation will be conducted at three assessment time points including baseline assessment (following initial medical intervention), assessment at the time of discharge from the intensive care center (ICU), and discharge from the hospital. After recruiting in this study, participants all receive the intervention of e-MCIT. If the subjects can complete the tasks, the results and completion times will be recorded. If the tasks cannot be completed, this situation and its probability will be documented as well. Due to the large number of measurement items in this study, it is expected to take a longer time. Breaks will be taken as needed according to each subject's tolerance. If the tasks cannot be completed in one session, they will be carried over to the next day. Our future study will be well-designed according to the result from this study.

Method: Patients with aSAH will be recruited, which Inclusion criteria for enrolment are as follows: (1) Diagnosis of spontaneous SAH resulting from aneurysm rupture confirmed by either CT scan or angiography. (2) Onset of stroke occurring in the acute phase, specifically 2-7 days after medical intervention. (3) Participants must be over 18 years old. (4) WFNS: 1-3. (5) Able to stand without support above 30 seconds. (6) Montreal Cognitive Assessment (MoCA)<26. Patients who present unstable vital sign (e.g., heart rate (HR): 40-100bpm, mean arterial pressure (MAP)> 80mmHg, respiratory rate (RR): 12-20, oxygen saturation (SpO2) > 95%, intracranial pressure (ICP) < 20mmHg and cerebral perfusion pressure (CPP) > 70mmHg) according to the criteria in previous study or evaluated as unsuitable by their attending physician will be excluded. Participants who are with other neurological disease might interfere the experiment and their education years less than 12 years will be excluded in this study. The e-MCIT consists of early mobilization and early cognitive training. Intervention will be 30 minutes per session, 4-5 sessions per week until discharging from the hospital. Outcome measurements includes side-effect events record, Montreal Cognitive Assessment (MoCA), Trail Making Test part A(TMT- A), Trail Making Test part B(TMT-B), Stroop color and word test (SCWT), forward and reverse digit span (DS) test, Go and no-go (GNG) test, Semantic Verbal Fluency test (SVFT), Fugl-Meyer Assessment for upper extremity (FMA- UE) and lower extremity (FMA-LE), Medical Research Council (MRC), Functional ambulatory category (FAC), kinematics performance in single and dual task ability, brain activity by functional Near-Infrared Spectroscopy (fNIRS) during all cognition assessment and in single and dual task, Functional independence measure (FIM), Modified Rankin Scale (mRS), Perme ICU mobility score, and National Institutes of Health Stroke Scale (NIHSS) . Statistical analysis was conducted using SPSS version 26.0. Categorical variables in the descriptive data of the participants were presented as numbers and percentages, while continuous variables were expressed as mean ± standard deviation. Nominal variables would be analyzed by X2 test. Wilcoxon Signed-Rank Test will be used to test the differences between pre-test and post-intervention time points due to small sample size. A two-tailed significance level (α) was set at 0.05. Thus, p< 0.05 revealed significant difference.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spontaneous SAH resulting from aneurysm rupture confirmed by either CT scan or angiography.
* Onset of stroke occurring in the acute phase, specifically 2-7 days after medical intervention.
* Participants must be over 18 years old.
* WFNS: 1-3.
* Able to stand without support above 30 seconds.
* Montreal Cognitive Assessment (MoCA)<26.

Exclusion Criteria:

* unstable vital sign (e.g., heart rate (HR): 40- 100bpm, mean arterial pressure (MAP)> 80mmHg, respiratory rate (RR): 12-20, oxygen saturation (SpO2) > 95%, intracranial pressure (ICP) < 20mmHg and cerebral perfusion pressure (CPP) > 70mmHg)
* patients evaluated as unsuitable by their attending physician
* those with other neurological diseases that might interfere with the experiment
* with less than 12 years of education

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Global cognition | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Global cognitive function will be measured by Montreal Cognitive Assessment (MoCA). Sum of score ranges from 0 to 30. There are eight subdivision of cognition category in this test, including visuospatial/ executive, naming, memory, attention, language, abstraction, delayed recall and orientation. Many studies assess global cognitive function in SAH patient by MoCA, which showed less ceiling or floor effect.
Executive function | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Executive function will be measured by three tests: Trail Making Test part A(TMT-A), Trail Making Test part B(TMT-B) and Stroop color and word test (SCWT), and scoring is based on time taken to complete the test with lower scores being better. Accuracy rate will be recorded as well.
Working memory | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Working memory will be measured by digit span (DS) test, which also usually represents subject's ability of verbal memory. Indicator for DS is the sum of the total scores for forward and reverse DS, with a score range of 0-30 points. A higher score indicates better performance.
Attention | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Attention ability will be measure by Go and no-go (GNG) test, which also represents subject's ability of set shifting, processing speed, and selective inhibition or also called inhibitory control.
Language ability | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  In category of language ability, verbal fluency will be measured by Semantic Verbal Fluency test (SVFT). The session consisted of three trials. Trials consisted of three different characters with the same pronunciation (20s / a Chinese character). The stimulation task was randomized to every subjects. Between three trails, there are 30 seconds in resting periods. Score 1 point for each correct answer, with total score of nine. Every correct and incorrect instance will be recorded. Accuracy rate (AR) will be calculated as the same method in GNG test. A higher accuracy rate also indicates better performance.

SECONDARY OUTCOMES:
Brain activity | T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Functional Near-Infrared Spectroscopy (fNIRS), which is a non-invasive neuro-imaging technique, will be used to detect the cerebral hemodynamics. The fNIRS data acquire via multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NYC, USA). Exports and receives dual-wavelength near-infrared signals are 760 and 850 nm. Data collection includes measurement changes in oxyhemoglobin [HbO], de-oxyhemoglobin [HbR] and the difference between HbO and HbR. The probe will not be placed above the surgical wound site. In cognition assessments: TMT-A& TMT-B, SCWT, DS, and GNG test, Optodes are configured to target both the bilateral prefrontal cortex (PFC) and the posterior parietal cortex (PPC). The setup involves 16 LED light sources and 16 detectors (16x16), resulting in 39 channels for the collection of hemodynamic data.
Motor impairment | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Motor impairment after stroke was measured by Fugl-Meyer Assessment for upper extremity (FMA-UE) and lower extremity (FMA-LE). In FMA-UE, part A to D, including subtests of upper extremity, wrist, hand, and coordination/ speed will be used only. The score ranges from 0 to 66. In FMA-LE, part E to F, including subtests of lower extremity, and coordination/ speed will be used only. The score ranges from 0 to 34. Both scores with higher score indicates better motor function
Muscle strength | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Key muscles strength was measured by Medical Research Council (MRC) scale. The scoring system is the same with manual muscle testing (MMT), with grade from 0 to 5. Total of score is 60, with higher scores indicating better strength.
Ability of ambulation | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Functional ambulatory category (FAC) would be used to assess the subject's ability of ambulation. FAC consists of six level, ranging from 0 to 5. The higher level indicates better ability of ambulation.
Functional Independence in ADL | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Functional independence measure (FIM) would be used to evaluate subject's ability of ADL. FIM consists of motor items and cognitive items.
  Motor items include subtest of self-care, sphincter control, mobility/ transfer, and locomotion. Cognitive items include subtest of communication and social cognition. The higher score indicates better independent ability. Scoring levels range from 1 to 7, thus, sum of score in FIM ranges from 18 to 126. The higher score indicates better independent ability.
Functional ability | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks), T2(discharge from hospital, an average of 4weeks)
  Modified Rankin Scale (mRS) would be used to assess the degree of disability or dependence in ADL. There are seven levels in mRS, with ranging from 0 to 6. Among this scale, the higher scale indicates less function ability.
Functional status in ICU | All tested at T0(baseline), T1(discharge from ICU, an average of 2 weeks)
  Perme ICU mobility score will be assessed at first time evaluation in ICU and discharge from ICU, which including mental status, potential mobility barriers, functional strength and functional ability. The higher score indicates better function status.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun R, Li X, Zhu Z, Li T, Li W, Huang P, Gong W. Effects of Combined Cognitive and Exercise Interventions on Poststroke Cognitive Function: A Systematic Review and Meta-Analysis. Biomed Res Int. 2021 Nov 17;2021:4558279. doi: 10.1155/2021/4558279. eCollection 2021. PMID 34840972
- [Background] Morello A, Spinello A, Staartjes VE, Bue EL, Garbossa D, Germans MR, Regli L, Serra C. Early versus delayed mobilization after aneurysmal subarachnoid hemorrhage: a systematic review and meta-analysis of efficacy and safety. Neurosurg Focus. 2023 Dec;55(6):E11. doi: 10.3171/2023.9.FOCUS23548. PMID 38262007
- [Background] Nussbaum ES, Mikoff N, Paranjape GS. Cognitive deficits among patients surviving aneurysmal subarachnoid hemorrhage. A contemporary systematic review. Br J Neurosurg. 2021 Aug;35(4):384-401. doi: 10.1080/02688697.2020.1859462. Epub 2020 Dec 21. PMID 33345644
- [Background] Geraghty JR, Lara-Angulo MN, Spegar M, Reeh J, Testai FD. Severe cognitive impairment in aneurysmal subarachnoid hemorrhage: Predictors and relationship to functional outcome. J Stroke Cerebrovasc Dis. 2020 Sep;29(9):105027. doi: 10.1016/j.jstrokecerebrovasdis.2020.105027. Epub 2020 Jun 20. PMID 32807442
- [Background] Karic T, Roe C, Nordenmark TH, Becker F, Sorteberg W, Sorteberg A. Effect of early mobilization and rehabilitation on complications in aneurysmal subarachnoid hemorrhage. J Neurosurg. 2017 Feb;126(2):518-526. doi: 10.3171/2015.12.JNS151744. Epub 2016 Apr 8. PMID 27058204